CLINICAL TRIAL: NCT05298800
Title: Clinical Observation of Combined Immunization of COVID-19 Inactivated Vaccine With Quadrivalent Influenza Vaccine(QIV) and 23-valent Pneumococcal Polysaccharide Vaccine
Brief Title: Combined Immunization of COVID-19 Inactivated Vaccine With QIV and PPV23
Acronym: QIV;PPV23
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Wu Jiang, Director，Head of the Institute for Vaccines and Immunization, Centers for Disease Control and Prevention, China
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BJCDCWJ202202
Record Dates: First submitted 2022-03-18; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Safety; Immunogenicity, Vaccine; COVID-19 Vaccines; Influenza Vaccines; Pneumococcal Vaccines
Keywords: Safety;Immunogenecity;Combined Immunization
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COVID-19 and QIV (Experimental)
  Interventions: Biological: Vaccine
- COVID-19 and PPV23 (Experimental)
  Interventions: Biological: Vaccine
- COVID-19 (Experimental)
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — Different arms were administrated different vaccines

SUMMARY:
The main objective of this study was to evaluate the immunogenicity and safety of the booster dose of COVID-19 inactivated vaccine and co-immunization with quadrivalent influenza vaccine and 23-valent pneumonia polysaccharide vaccine in people aged 18 years and older. A randomized controlled, open trial design was adopted.

The study was conducted with informed consent of the subjects for immunogenicity and safety in the population aged 18 years and older. A total of 3000 healthy subjects were selected, (1)600 healthy subjects were selected for the immunogenicity and safety study of co-immunization, 300 in the adult group (18-59 years old) and 300 in the elderly group (60 years old and above); (2) 2400 healthy subjects were selected for the observational study of the safety of co-immunization, 1200 in the adult group (18-59 years old) and 1200 in the elderly group (60 years old and above ) 1200 people.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18 years old and older
* Over 6 months after primary immunization with COVID-19 vaccines
* Can understand and sign the consent
* Can provide effective personal identification

Exclusion Criteria:

* Has a history of COVID-19 infection
* Less than 6 months after primary immunization with COVID-19 vaccines
* Already vaccinated with influenza vaccines of that year
* Vaccinated with pneumococcal vaccines within 5 years
* Has a history of severe hypersensitivity reaction to vaccines
* Has uncontrolled seizure or other severe neural system illnesses
* Has a fever, chronic disease, or acute disease during immunization
* Gestation period, lactation period, or planning to get pregnant within 3 months
* Administrated with other drugs under research within 30 days before vaccination
* Received attenuated vaccines within 14 days before vaccination
* Received subunit vaccines or inactivated vaccines within 7 days before vaccination
* Other conditions based on researcher's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate of neutralizing antibody | 28 days after the third dose of COVID-19 vaccine

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Daxing District Center of Disease Control and Prevention, Beijing
  - Huairou District Center of Disease Control and Prevention, Beijing
  - Miyun District Center of Disease Control and Prevention, Beijing

REFERENCES:
- [Derived] Bai S, Zhou S, Zhang J, Chen W, Lv M, Wang J, Zhang A, Wu J, Zhao W. Immunogenicity and safety of different combinations involving a third booster dose of SARS-CoV-2 inactivated vaccine, inactivated quadrivalent influenza vaccine, and 23-valent pneumococcal polysaccharide vaccine in adults aged >/=60 years: a phase 4, randomized, open-label study. Front Immunol. 2024 Aug 20;15:1437267. doi: 10.3389/fimmu.2024.1437267. eCollection 2024. PMID 39229259
- [Derived] Zhou S, Lv M, Bai S, Chen W, Zhao W, Wang J, Zhang A, Li J, Xie H, Gao Y, Li D, Wu J. Baseline Pneumococcal IgG Levels and Response to 23-Valent Pneumococcal Polysaccharide Vaccine among Adults from Beijing, China. Vaccines (Basel). 2023 Nov 29;11(12):1780. doi: 10.3390/vaccines11121780. PMID 38140184